CLINICAL TRIAL: NCT05433220
Title: PRagmatic Trial Of Messaging to Providers About Treatment of Heart Failure (PROMPT-HF) at Inova
Brief Title: PRagmatic Trial Of Messaging to Providers About Treatment of Heart Failure at Inova
Acronym: PROMPTHF-Inova
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: U22-04-4736
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure
Keywords: Heart Failure; GDMT; NYHA; HFrEF; Implementation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alert when provider is entering orders (Experimental)
  Interventions: Other: Best Practice Advisory using Electronic Health Record
- No alert, usual care (No Intervention)

INTERVENTIONS:
Other: Best Practice Advisory using Electronic Health Record — Providers caring for patients randomized to the intervention arm will have a best practice alert appear for each of their eligible patients upon opening of the order entry screen in the patient's medical record. This alert informs the provider to the presence of HFrEF, notes the patient's current LVEF and current evidence-based medications, and gives access to an order set with recommended evidence- based, guideline-recommended, and FDA- approved therapies for patients with HFrEF. Providers will also have access to a link to best available guideline recommended information regarding treatment of heart failure to allow further education if desired by the provider. The alerts will also clearly state the expected monitoring and follow-up required for prescriptions of these medications.
  Arms: Alert when provider is entering orders

SUMMARY:
A randomized, single-blind intervention trial to test the comparative effectiveness of an electronic health record best practice advisory system that informs clinicians of guideline-indicated and FDA-approved heart failure medications currently not prescribed to their patients with heart failure versus usual care (no alert and how things are done currently). The purpose of the alert is to stimulate appropriate medication prescription for patients with heart failure and a reduced ejection fraction. This will be done across outpatient Inova clinics and at the five Inova hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 Years
* Seen by a Cardiologist in an Inova clinic or Inova hospital setting
* Left Ventricular Ejection Fraction ≤40%

Exclusion Criteria:

* Opted out of EHR-based research
* Hospice care
* Already receiving maximally titrated doses of each of the four classes of evidence- based HFrEF medical therapy
* Prior heart transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2022-08-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Increased use of GDMT in patients with Heart Failure with Reduced Ejection Fraction | 30 days after randomization
  The primary outcome for the trial will be the proportion of patients with HFrEF who have an increase in the number of prescribed evidence-based therapies for HFrEF (beta-blockers, ACE-I/ARB/ARNI, MRA, SGLT2i) 30 days after randomization.

SECONDARY OUTCOMES:
All-cause hospitalization and all-cause mortality at 30 days | 30 days
  Outcomes will be determined by review of medical, hospital, and billing records.
All-cause hospitalization and all-cause mortality at 90 days | 90 days
  Outcomes will be determined by review of medical, hospital, and billing records.
All-cause hospitalization and all-cause mortality at 180 days | 180 days
  Outcomes will be determined by review of medical, hospital, and billing records.
All-cause hospitalization and all-cause mortality at 1 year | 1 year
  Outcomes will be determined by review of medical, hospital, and billing records.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Psotka, MD, PhD, Principal Investigator — Inova Health Care Services
Locations (1):
- Inova Health System, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Only aggregate participant data will be reported upon the completion of the project.

REFERENCES:
- See also: PRagmatic Trial Of Messaging to Providers About Treatment of Heart Failure in the Inpatient Setting (PROMPT-HF) — https://clinicaltrials.gov/ct2/show/NCT04686604?term=PROMPT-HF&draw=2&rank=1